CLINICAL TRIAL: NCT02080156
Title: Impact of Continuous Positive Airway Pressure Therapy on Outcomes in Patients Undergoing Coronary Revascularization
Brief Title: Impact of Continuous Positive Airway Pressure (CPAP) Therapy on Outcomes in Patients Undergoing Coronary Revascularization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Xiandao Yuan M.D., MD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMU-881206
Record Dates: First submitted 2014-02-22; First posted 2014-03-06 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Obstructive Sleep Apnea; Ischaemic Heart Desease
Keywords: Obstructive Sleep Apnea; Percutaneous Coronary Intervention; Coronary Artery Bypass Graft; Mortality; Questionnaire; Biomarker
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no-CPAP (No Intervention): CPAP vs. no-CPAP in patients undergoing Coronary Revascularization follow-up for 3 years
- CPAP (Experimental): CPAP vs. no-CPAP in patients undergoing Coronary Revascularization follow-up for 3 years
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP
  Arms: CPAP

SUMMARY:
Investigators assume that continuous positive airway pressure (CPAP) therapy can reduce the mortality, stroke rate and secondary coronary surgery in CAD with obstructive sleep apnea (OSA) patients after percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABA) during postoperative follow-up of 3 years.

DETAILED DESCRIPTION:
Investigators observe whether continuous positive airway pressure (CPAP) therapy can reduce the mortality, stroke rate and secondary coronary surgery in CAD with OSA patients after percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABA) during postoperative follow-up of 3 years. During the 3 years, we randomize all enrolled patients to 2 groups separately beginning CPAP or no-CPAP intervention after sleep monitoring. Guidance for all patients during follow-up 1 week, 2 week, 1 month, 3 month. The follow-up procedure includes clinical assessments at three months, six months, one year, two and three years respectively.The primary outcome variables are prospectively being documented and are not subject to observer bias.Baseline comorbidity data, results of the sleep recordings, compliance with CPAP device, scores of the questionnaires as well as results of the blood analysis are performed and/or documented consecutively in separate files by research personnel blinded to the allocation of the study groups and/or unaware of the results of the concomitant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Angiography confirmed coronary heart disease (CHD) patients
* Underwent PCI or coronary artery bypass graft (CABG) in recent the week
* Signed informed consent
* Mild-to-moderate OSA（5≤AHI≤100)

Exclusion Criteria:

* OSA patients who has already started treatment
* Patients presenting mainly central apnea (≥ 50%)
* Respiratory insufficiency patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yongxiang Wei, MD PhD, Study Chair — Capital Medical University Affiliated Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China